CLINICAL TRIAL: NCT03846648
Title: A Randomized, Placebo-controlled, Double-blind Phase I Study to Explore Safety, Tolerability and Pharmacodynamics of CyPep-1 in Subjects With Cutaneous Warts
Brief Title: CyPep-1 in Cutaneous Warts
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre for Human Drug Research, Netherlands (Other)
Responsible Party: Principal Investigator, Clintrials CHDR, PhD, Centre for Human Drug Research, Netherlands
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHDR1803; NL67664.056.18 (Other: ToetsingOnline CCMO)
Record Dates: First submitted 2019-01-25; First posted 2019-02-19 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Cutaneous Warts

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blind phase I study
Who Masked: Participant, Investigator
Masking Description: This study will be performed in a double-blind fashion. The investigator, study staff, subjects, sponsor, and monitor will remain blinded to the treatment until study closure. The investigational drug and its matching placebo are indistinguishable and will be packaged in the same way.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cypep-1 (Active Comparator): CyPep-1 cream 1% (w/w) will be applied once daily on a 5x5 cm healthy skin area on the upper back and on 1 to max 3 common warts on the (dorsal/palmar) side of the hand.
  In Part 1 the dosing will be performed once daily for 7 days. The dose of 200 μL CyPep-1 cream will be applied on a 5x5 cm on the back by clinical staff. In addition, up to 3 common warts will be treated with 20 μL of the CyPep1 cream per day.
  In Part 2 subjects will administer 20-30 mg CyPep-1 cream once daily at home after instruction by clinical staff. The total treatment period will be 28 days, possibility of a maximum extension of three days is allowed.
  Interventions: Drug: Cypep-1
- Placebo (Placebo Comparator): Placebo cream (the same as that of the drug product CyPep-1 1% (w/w) but without the active substance) will be applied once daily on the same areas as described above.
  Interventions: Drug: Cypep-1

INTERVENTIONS:
Drug: Cypep-1 — Eligible subjects will be randomized to one of the two treatment groups in a ratio of 1:1 (active:placebo).
  The treatment groups are:
  * CyPep-1 topical formulation 1% (w/w)
  * Vehicle topical formulation (placebo) The minimum set of studied warts is 1 treated common wart per subject. The subjects will be randomly assigned to treatment. During the treatment period topical formulation will be applied daily on to a maximum of 3 warts. One selected wart will serve as target wart, i.e. the primary wart, for detailed analysis. Selection of warts will be based on the feasibility to conduct treatment application and pharmacodynamics (including biopsy sampling) on the region of interest.

SUMMARY:
This Phase 1 study is intended to explore the safety, tolerability, pharmacodynamics and efficacy of topical CyPep-1 as a potential treatment for HPV-associated conditions. Since this is a first-on-human study of a topical formulation, the first subjects will be monitored more frequently in order to establish the safety profile. Because clinical outcomes (i.e. reduction/clearance of the lesion) often require lengthy treatment / observation periods, the study design will primarily utilize clinical measurements of wart dimensions, along with HPV viral load as a biomarker of anti-viral effect.

DETAILED DESCRIPTION:
This study has a phase 1, randomized, vehicle-controlled, double-blind, single center design to explore the safety, tolerability and pharmacodynamics (PD) of topically applied CyPep-1 in otherwise healthy patients with cutaneous warts.

The study will entail two parts. Part 1 will follow a target area of 5x5 cm healthy skin to study tolerability and safety of the formulation. During this study part also a maximum of 3 common warts, preferably at the dorsal or palmar side of the hand / finger(s), will be treated. Several assessments will be done to determine pharmacodynamics and to explore possible efficacy after a treatment period of 1 week.

Part 2 will evaluate the pharmacodynamics and efficacy of CyPep-1 after a treatment period of 4 weeks. Study part 2 will commence after an interim analysis, e.g. a blind data review, of study part 1 has been conducted.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects (male, non-pregnant female), 18 to 65 years of age, inclusive. (Healthy status is defined by absence of evidence of any clinical significant/uncontrolled active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs,12-lead ECG, haematology, blood chemistry, and urinalysis);
* Body mass index (BMI) between 18 and 35 kg/m2, inclusive;
* Free of clinically significant systemic or dermatologic disorders, which, in the opinion of the investigator, will interfere with the study results or increase the risk of Adverse Events;
* Have at least 1 (non-peri/subungual) common wart on the, preferably, dorsal/palmar side of the hand / fingers which is 3-10 mm (inclusive) in diameter in its longest dimension on the plane of the skin;
* If female of childbearing potential, have a negative urine pregnancy test at Screening/Day 0, and are willing to use effective contraception during the study (i.e. oral, implanted, injectable, IUD, diaphragm, condom, tubal ligation, abstinence, or are in a monogamous relationship with a partner who has had a vasectomy);
* Able to participate and willing to give written informed consent and to comply with the study restrictions;
* Ability to communicate well with the investigator in the Dutch language;
* Willing to refrain from using cosmetics or other topical products in the treatment area for the duration of the study;
* Agree not to use wart-removing products (prescription or over-the-counter) in the target area or prohibited medications other than the study medication during the course of the study.

Exclusion Criteria:

* Any clinically significant abnormality as determined by medical history taking and physical examinations obtained during the screening visit that in the opinion of the investigator would interfere with the study objectives or compromise subject safety;
* Not willing to use effective (double barrier) contraception until at least 3 months after last study drug application;
* For women: a positive pregnancy test and/or breastfeeding at screening or women who plan to become pregnant;
* A positive test for drugs of abuse at screening;
* History of alcohol or illicit drug abuse (alcohol abuse defined as alcohol consumption > 21 units/week);
* Positive test results for Hepatitis B, Hepatitis C or HIV;
* Have used salicylic acid or any other over-the-counter wart-removing product including cryotherapy in the treatment area within 28 days prior to first study drug application;
* Have required systemic intake of immunosuppressive or immunomodulatory medication (including oral or parenteral corticosteroids) within 60 days prior to first study drug application or during the course of the study. Routine use of inhaled or intranasal corticosteroids during the study is allowed;
* Have any current and / or recurrent clinical significant skin infection in the treatment area other than common warts;
* Have a known sensitivity to any of the investigational product ingredients;
* Participation in an investigational drug or device study within 3 months prior to screening or more than 4 times in the past year;
* Donation of blood or blood loss of >500 mL within 3 months prior to screening or donation of plasma within 14 days
* Not having a general practitioner;
* Not willing to give permission to have the general practitioner to be notified upon participation in this study;
* Any condition that in the opinion of the investigator would complicate or compromise the study or the well-being of the subject.

Part 2 only:

- Have treatment resistant / persistent warts as defined as one of the following:

1. More than 5 different failed treatments including topical formulations and cryotherapy
2. Longer than 6 years presence of the target wart
3. Having received active treatment in a clinical trial with an experimental drug for cutaneous warts.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Changes in heart rate | Part 1: Baseline, 0.5h, 2h, 4h, 8h, 24h, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 14, Day 21. Part 2: All study visits.
  Part 1:
  Heart rate (number of pulses/min) will be measured during the time points described below.
Changes in blood pressure (systolic and diastolic) | Part 1: Baseline, 0.5h, 2h, 4h, 8h, 24h, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 14, Day 21. Part 2: All study visits.
  Blood pressure (mmHg) will be measured during the time points described below.
Changes in body temperature | Part 1: Baseline, 0.5h, 2h, 4h, 8h, 24h, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 14, Day 21. Part 2: All study visits.
  Body temperature (degrees Celsius) will be measured during the time points described below.
Recording of (S)AEs | At all study visits.
  AEs and AEs will be recorded during all visits.

SECONDARY OUTCOMES:
Changes in wart size | Part 1: Baseline, 24h,Day 3, Day 5, Day 7, Day, 14 and Day 21, Part 2: all study visits
  Wart size (in mm) will be measured during the time points described below.
HPV viral load | 24-48h during Part 1, 1-6 weeks during Part 1 and Part 2
  Part 1:
  Swabs will be obtained every 48h during treatment period and at the FU visits.
  Part 2:
  Swabs will be obtained at all study visits.

OTHER OUTCOMES:
Pharmacokinetics of CyPep-1 | 24h during Part 1, Day 14 during Part 1 and Day 28 during Part 2.
  Blood samples will be collected for measurement of CyPep-1 plasma concentration.
  Part 1:
  Daily during treatment period and at Day 14.
  Part 2:
  At Day 28 (End of Trial)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Human Drug Research, Leiden, South Holland, Netherlands